CLINICAL TRIAL: NCT05904678
Title: Anatomical and Functional Assessment of Ex-vivo Coronary Perfusion
Acronym: ECHORONEX
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-A02579-32
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Cardiac Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Heart transplantation is the gold standard treatment for advanced heart failure, with a survival rate >60% at 10 years. Heart transplantation activity has tended to decline significantly in France since 2017, with -5% of transplants per year according to the Agence de la Biomédecine report (La Plaine-Saint-Denis, France, https://rams.agence-biomedecine.fr). Graft selection criteria have been extended over the past two decades, in particular the average donor age, which currently exceeds 50 in France. These donors with extended criteria are more exposed to the risk of acquired coronary lesions. The current indications for donor coronary angiography are age >55 or >45 with at least two cardiovascular risk factors, but it is performed in only a third of these cases. Coronary angiography would increase the chances of graft acceptance by 9%.

At the same time, some heart transplants are rejected for lack of a complete functional evaluation, or because they present moderate left ventricular dysfunction. In catecholaminergic stress cardiomyopathy, left ventricular dysfunction is reversible, but its recovery kinetics are difficult to predict. Ex vivo resuscitation of these grafts on a perfusion machine could enable functional recovery and acceptance of these grafts for transplantation. This approach could also be applied to other cardiac grafts harvested from donors with extended criteria, such as prolonged cardiac arrest.

Graft preservation on ex vivo perfusion machines has enjoyed considerable growth over the past decade. The Organ Care System (OCS, TransMedics, Andover, USA) is currently the only transportable perfusion machine available and marketed for clinical use, with experience of over 1,000 transplants worldwide. OCS technology is based on isolated ex vivo perfusion of the heart with normothermic blood in Langendorff mode (retrograde aortic perfusion). This transportable platform enables metabolic evaluation of the graft based on the concentration of circulating lactate in the perfusate, a criterion of viability and "transplantability". The aims of this alternative method to static hypothermic preservation of heart grafts are threefold: 1) to extend the preservation time of the heart graft; 2) to assess graft viability prior to transplantation; 3) to resuscitate a heart graft harvested after controlled circulatory arrest (Maastricht 3).

Since February 2019, 31 heart grafts have been placed on OCS in France thanks to the implementation of an ex vivo perfusion program at the Lille and Rennes teaching hospitals, and the Marie Lannelongue Hospital. Our preliminary results have recently been accepted for publication. In this research project, we propose to analyze in real time the quality of coronary perfusion using vasculoscopy on isolated human hearts placed on OCS, and to put this anatomical and functional assessment into perspective with the results of heart transplantation.

Indeed, vasculoscopy is an innovative non-invasive imaging approach that has never before been applied in the cardiovascular field. We aim to validate this technology in the assessment of myocardial perfusion quality of the machine-perfused graft awaiting transplantation, by correlating the signal obtained with perfusion parameters on OCS (coronary flow, mean aortic pressure, arterial and venous lactate) as well as with transplant outcomes (primary graft failure rate, recipient survival rate at one month post-transplant). Myocardial perfusion parameters have never been correlated with heart transplantation outcomes to date.

ELIGIBILITY:
Inclusion Criteria:

- Adult patient going for heart transplantation with cardiac transplantation on ex vivo perfusion machine.

Exclusion Criteria:

* Patient opposing study participation.
* Minor patient

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient going for heart transplantation with cardiac transplantation
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-11-15 (Estimated); Study Completion 2024-02-15 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of coronary lesions identified by vasculoscopy | 1 DAY

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No